CLINICAL TRIAL: NCT06243705
Title: Assessing the Effectiveness of Robot-pets in Reducing Dental Anxiety in Children: A Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Robot-pets in Reducing Dental Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Melis AKYILDIZ, Post Doctoral Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ADUDHF-2023/23
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Dental Anxiety
Keywords: Behaviour management; Robot pet; Dental anxiety

STUDY DESIGN:
Intervention Model Description: The study will be used a parallel-group randomized controlled trial design. Children fulfilling the inclusion criteria will be randomized to three group. Fissure sealants will be applied to the children using the distraction technique determined by randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot-Pet Group (Experimental): The robot-pet sits on the child's lap while the fissure sealant is applied. Preoperative (T1) baseline levels of dental anxiety will be measured using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) and the Facial Image Scale (FIS), and behavior rating will be measured using the Frankl Behavior Rating Scale (FBRS). Intraoperative (T2) cooperation level will be recorded using the Modified Houpt Scale (MHS) during the surface cleaning (T2A), isolation (T2B) and washing (T2C) phases of fissure sealant application. Postoperative(T3) anxiety level and behavior rating measurements (CFSS-DS, FIS, FBRS) will be repeated. Physiological markers for dental anxiety, such as heart rate and oxygen saturation, will be measured at all time points (T1, T2A-B-C, T3). Children and parents in this group will received a questionnaire for their perception about the use of their distraction technique(T3).
  Interventions: Device: Robot-Pet
- Virtual Reality Glasses Group (Active Comparator): During the application of fissure sealant, the child watches a cartoon through virtual reality glasses. Preoperative (T1) baseline levels of dental anxiety will be measured using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) and the Facial Image Scale (FIS), and behavior rating will be measured using the Frankl Behavior Rating Scale (FBRS). Intraoperative (T2) cooperation level will be recorded using the Modified Houpt Scale (MHS) during the surface cleaning (T2A), isolation (T2B) and washing (T2C) phases of fissure sealant application. Postoperative(T3) anxiety level and behavior rating measurements (CFSS-DS, FIS, FBRS) will be repeated. Physiological markers for dental anxiety, such as heart rate and oxygen saturation, will be measured at all time points (T1, T2A-B-C, T3). Children and parents in this group will received a questionnaire for their perception about the use of their distraction technique(T3).
  Interventions: Device: Virtual Reality Glasses
- Control Group (No Intervention): Tell-Show-Do technique will be used to apply the fissure sealant. No additional distraction will be applied. Preoperative (T1) baseline levels of dental anxiety will be measured using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) and the Facial Image Scale (FIS), and behavior rating will be measured using the Frankl Behavior Rating Scale (FBRS). Intraoperative (T2) cooperation level will be recorded using the Modified Houpt Scale (MHS) during the surface cleaning (T2A), isolation (T2B) and washing (T2C) phases of fissure sealant application. Postoperative(T3) anxiety level and behavior rating measurements (CFSS-DS, FIS, FBRS) will be repeated. Physiological markers for dental anxiety, such as heart rate and oxygen saturation, will be measured at all time points (T1, T2A-B-C, T3).

INTERVENTIONS:
Device: Robot-Pet — The robot-pet makes sounds like a real cat and responds to touch and petting
  Arms: Robot-Pet Group
Device: Virtual Reality Glasses — VR glasses allow you to see videos and films projected on the screen more realistic. With its filtering feature, it combines two different images in the brain and provides the perception of depth in the image and creates a 3D space environment
  Arms: Virtual Reality Glasses Group

SUMMARY:
Dental anxiety is a psychological condition marked by fear and worry about potential negative experiences during dental treatment, often accompanied by a feeling of loss of control. Dental anxiety is common in children and adolescents and is associated with a lower quality of life related to oral health. Furthermore, it correlates with an increased incidence of untreated caries. Using behavioral management techniques can help children cope with dental anxiety, making it easier for them to undergo treatment in a positive and healthy way.

Primarily aim of this study is to evaluate the effectiveness of using a robot-pet to reduce dental anxiety in children. Additionally, the research aims to compare the efficacy of this technique with the audiovisual distraction technique and to evaluate children's perceptions regarding the use of a robot-pet.

DETAILED DESCRIPTION:
Dental anxiety is a universal phenomenon that affects people of all ages in different countries. This condition negatively affects the quality of life related to oral health in children and adults. Dental anxiety has a negative impact on children's oral and dental health. Studies have reported that children with dental anxiety have poorer oral hygiene and untreated dental caries.

Basic behavior management strategies are commonly employed in dental offices to shape a child's behavior, teach coping skills, instill positive attitudes, build trust, and enable effective and efficient treatment. These strategies include traditional techniques such as tell-show-do and voice control, as well as contemporary techniques such as cognitive behavioral therapy and audio-visual distraction.

Tell-Show-Do (TSD) is a well-known basic behavioral technique. This technique involves verbally explaining dental procedures or instruments to the child using developmentally appropriate language. The visual, auditory, olfactory, and tactile aspects of the procedure are then demonstrated to the patient in a carefully defined, non-threatening environment. Finally, the procedure is performed without deviating from the initial explanation and demonstration.

Audiovisual distraction is a technique that combines visual and auditory components. It involves a spectacle system that consists of a head-mounted display and in-ear headphones. The aim is to reduce visual and auditory interference from the sounds and images of the dental working environment. This technique is intended to distract children during dental treatment by immersing them in a two- or three-dimensional world. According to some suggestions, this application may be more effective than traditional distraction methods due to its technological and engaging nature.

Animal-assisted therapy is a targeted intervention that uses a trained animal in a healthcare setting to improve patient interactions or reduce anxiety, pain, or distress. Appointments for animal-assisted therapy are scheduled for a specific time and duration, and the animals used have undergone temperament testing, rigorous training, and certification. According to a report, animals used during dental visits can help patients overcome communication barriers and reduce stress related to treatment by establishing a safe and relaxing relationship with the dentist. Animal-assisted therapies can increase children's compliance in the clinic and distract their attention. However, due to clinical hygiene conditions, it may pose risks to both trained animals and dental personnel. If necessary, precautions are taken, it can be applied. To eliminate the mentioned risks and difficulties, robots in cat/dog form can be used to apply this useful technique. In this context, it is important to keep up with developments in behavior management and assess their suitability for clinical practice. It is believed that using a robot-pet can enhance children's cooperation during dental procedures. This study provides guidance for clinicians on an alternative method of behavior management.

Methods:

A total of 72 children aged 6-10 years with no previous dental experience, needs fissure sealant treatment will be included in this study. Children will be randomly assigned to three groups according to received distraction technique during fissure sealant application; each group having 24 patients as follows: Group-1: Robot-Pet, Group-2:Virtual Reality Glasses, and Group 3: Tell-Show-Do (Control). Anxiety levels and behaviors will be assessed at different timepoints. Preoperative (T1) baseline levels of dental anxiety will be measured using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) and the Facial Image Scale (FIS), and behavior rating will be measured using the Frankl Behavior Rating Scale (FBRS). Intraoperative (T2) cooperation level will be recorded using the Modified Houpt Scale (MHS) during the surface cleaning (T2A), isolation (T2B) and washing (T2C) phases of fissure sealant application. Postoperative(T3) anxiety level and behavior rating measurements (CFSS-DS, FIS, FBRS) will be repeated. Physiological markers for dental anxiety, such as heart rate and oxygen saturation, will be measured at all time points (T1, T2A-B-C, T3). An independent evaluator, who will have been formally trained regarding the two behavior scales(FBRS,MHS), will observe and record all data. Children and parents in the Group 1 and 2 will received a questionnaire for their perception about the use of their distraction technique(T3).

Statistical Analyses:

The IBM SPSS Statistics for Windows, Version 25.0 (Released 2017, Armonk, NY: IBM Corp.) package program will be used for statistical analyses. Numeric variables without an issue of normal distribution fit will be compared among three groups using the One-Way Analysis of Variance (ANOVA) method. In cases where homogeneity is not established, the Welch Test will be employed for multiple comparisons, and Dunnett's T3 method for pairwise comparisons.All hypothesis tests will be conducted at a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria: : Children are eligible for inclusion if;

* They are 6 to 10 years old
* They have no previous dental treatment
* They have at least one of the permanent first molars is fully erupted

Exclusion Criteria: Children will be excluded from the study if;

* They do not have a parental agreement to participate
* They need emergency care, such as dental trauma or pain
* They have incomplete eruption of all permanent first molars
* They have special health care needs, intellectual disabilities or autism spectrum disorders
* They have phobia of animals such as cats or dogs
* If their Frankl Behaviour Rating Score is 1 (Strongly Negative)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Assesment of Heart Rate and Oxygen Saturations | Before Treatment, During Fissure Sealant Application-Surface Cleaning Phase, During Fissure Sealant Application-Isolation Phase, During Fissure Sealant Application-Washing Phase, Immediately After Treatment
  Evaluation of the physiological parameters heart rate and oxygen saturation shows the interaction between the autonomic nervous system and dental anxiety. These values provide information about the children's cardiovascular and respiratory responses during treatment.
Assesment of Behaviour- Frankl Behaviour Rating Scale | Before Treatment, Immediately After Treatment
  Dental professionals uses this scale to systematically assess and record information about child's behaviour in the dental clinic environment.The behaviour is rated from 1 to 4 (strongly negative (1), negative (2), positive (3), strongly positive (4))
Assesment Of Behaviour- Modified Houpt Behaviour Rating Scale | During Fissure Sealant Application-Surface Cleaning Phase, During Fissure Sealant Application-Isolation Phase, During Fissure Sealant Application-Washing Phase
  This is a three-stage scale designed to assess the child's compliance and cooperative behaviour during dental treatment. It is a scale in which the child is assessed by the dental practitioner on three different parameters relating to movement, crying and overall behaviour and scored from 1 to 4 according to their behaviour.
  Movement: 1=no movement 2= Controllable movement 3=Continuous movement 4=Violent movement Crying: 1= No crying 2= Intermittent mild crying 3= Continuous persistent crying 4= Hysterical crying Overall Behaviour: 1= Excellent, treatment completed 2= air, treatment interrupted, but eventually all completed 3= oor, treatment interrupted, only partial treatment completed 4= Aborted, no treatment rendered
Assesment of Dental Anxiety- Children's Fear Survey Schedule-Dental Subscale | Before Treatment, Immediately After Treatment
  The Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) is a specific tool designed to assess dental anxiety and fear in children.
  1. Dentists
  2. Doctors
  3. Injections
  4. Having somebody examine your mouth
  5. Having to open your mouth
  6. Having a stranger touch you
  7. Having somebody look at you
  8. The dentist drilling.
  9. The sight of the dentist drilling
  10. The noise of the dentist drilling
  11. Having somebody put instruments in your mouth
  12. Choking
  13. Having to go to the hospital
  14. People in white uniforms
  15. Having the dentist clean your teeth Each item was scored between 1-5 according to the answer given (Scoring is as follows: 1= Not afraid at all, 2= A little afraid, 3= Moderately afraid, 4= Quite afraid, 5= Very afraid).
Assesment of Dental Anxiety- Facial Image Scale | Before Treatment, Immediately After Treatment
  The Facial Image Scale consists of a series of five faces ranging from very happy to very unhappy. Children were asked to point to which face they felt most like at that moment. The scale is scored by rating the face with the most positive affect as 1(Very Happy) and the face with the most negative affect as 5(Very Unhappy).

SECONDARY OUTCOMES:
Evaluate the Child's Perspectives on the Use of Robot-Pet | Immediately After Treatment
  A questionnaire will be carried out through an interview with children to determine what their perception of robot-pet.
  1. I liked having a robot cat on my lap.
  2. It felt good to be treated with a robot cat on my lap.
  3. Dental treatments are easier when I have a robot cat on my lap.
  4. I will tell my friends that I have been treated with a robot cat.
  5. I would have the treatment even if I did not have a robot cat on my lap. The scale is 1 (strongly agree) 2 (agree) 4 (no opinion) 4 (disagree) 5 (strongly disagree) A higher score indicates a worse outcome.
Assesment of Parents' Perspectives on the Use of Robot-Pet | Immediately After Treatment
  A questionnaire will be carried out through an interview with parents to determine what their perception of robot-pet.
  1. Treatment with robot cat helped my child cope with dental anxiety.
  2. I would recommend treatment with a robot cat to others.. The scale is 1 (strongly agree) 2 (agree) 4 (no opinion) 4 (disagree) 5 (strongly disagree) A higher score indicates a worse outcome.
Evaluate the Child's Perspectives on the Use of Virtual Reality Glasses | Immediately After Treatment
  A questionnaire will be carried out through an interview with children to determine what their perception of virtual reality glasses.
  1. I liked watching cartoons with glasses.
  2. It felt good to be treated while watching cartoons with glasses.
  3. Dental treatment will be easier when I watch cartoons with glasses.
  4. I will tell my friends that I was treated by watching cartoons with glasses.
  5. Even if I didn't watch cartoons with glasses, I would have the treatment. The scale is 1 (strongly agree) 2 (agree) 4 (no opinion) 4 (disagree) 5 (strongly disagree) A higher score indicates a worse outcome.
Assesment of Parents' Perspectives on the use Virtual Reality Glasses | Immediately After Treatment
  A questionnaire will be carried out through an interview with parents to determine what their perception of virtual reality glasses.
  1. Treatment with virtual reality glasses helped my child cope with dental anxiety.
  2. I would recommend treatment with virtual reality glasses to others. The scale is 1 (strongly agree) 2 (agree) 4 (no opinion) 4 (disagree) 5 (strongly disagree) A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Melis AKYILDIZ, PhD, Study Director — Aydin Adnan Menderes University
Locations (1):
- Melis AKYILDIZ, Aydin, Efeler, Turkey (Türkiye)

REFERENCES:
- [Background] Gilchrist F, Campbell C. Communication and the Use of Language. In: Dental Fear and Anxiety in Pediatric Patients. Cham: Springer International Publishing; 2017. p. 117-36.
- [Background] Gilchrist F, Marshman Z, Deery C, Rodd HD. The impact of dental caries on children and young people: what they have to say? Int J Paediatr Dent. 2015 Sep;25(5):327-38. doi: 10.1111/ipd.12186. Epub 2015 Jul 8. PMID 26153526
- [Background] Alsadat FA, El-Housseiny AA, Alamoudi NM, Elderwi DA, Ainosa AM, Dardeer FM. Dental fear in primary school children and its relation to dental caries. Niger J Clin Pract. 2018 Nov;21(11):1454-1460. doi: 10.4103/njcp.njcp_160_18. PMID 30417844
- [Background] Akbay Oba A, Dulgergil CT, Sonmez IS. Prevalence of dental anxiety in 7- to 11-year-old children and its relationship to dental caries. Med Princ Pract. 2009;18(6):453-7. doi: 10.1159/000235894. Epub 2009 Sep 30. PMID 19797921
- [Background] Wigen TI, Skaret E, Wang NJ. Dental avoidance behaviour in parent and child as risk indicators for caries in 5-year-old children. Int J Paediatr Dent. 2009 Nov;19(6):431-7. doi: 10.1111/j.1365-263X.2009.01014.x. Epub 2009 Aug 25. PMID 19708863
- [Background] Shim YS, Kim AH, Jeon EY, An SY. Dental fear & anxiety and dental pain in children and adolescents; a systemic review. J Dent Anesth Pain Med. 2015 Jun;15(2):53-61. doi: 10.17245/jdapm.2015.15.2.53. Epub 2015 Jun 30. PMID 28879259
- [Background] American Academy of Pediatric Dentistry. Behavior guidance for the pediatric dental patient. The Reference Manual of Pediatric Dentistry. Chicago, Ill.: American Academy of Pediatric Dentistry; 2023:359-77.
- [Background] Liu Y, Gu Z, Wang Y, Wu Q, Chen V, Xu X, Zhou X. Effect of audiovisual distraction on the management of dental anxiety in children: A systematic review. Int J Paediatr Dent. 2019 Jan;29(1):14-21. doi: 10.1111/ipd.12430. Epub 2018 Oct 26. PMID 30362187
- [Background] Charowski M, Wells MH, Dormois L, Fernandez JA, Scarbecz M, Maclin M. A Randomized Controlled Pilot Study Examining Effects of Animal Assisted Therapy in Children Undergoing Sealant Placement. Pediatr Dent. 2021 Jan 15;43(1):10-16. PMID 33662243